CLINICAL TRIAL: NCT00165737
Title: A 24-Week, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Evaluation of the Efficacy, Safety and Tolerability of Donepezil Hydrochloride (E2020) in Patients With Dementia Associated With Cerebrovascular Disease
Brief Title: Donepezil Hydrochloride (E2020) in Dementia Associated With Cerebrovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Margaret Moline, Ph.D, Study Director, Eisai Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-319
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Dementia, Vascular
Keywords: Dementia cerebrovascular disease
MeSH Terms: conditions — Dementia, Vascular | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Donepezil Hydrochloride

SUMMARY:
Twenty-four week, prospective, randomized, double-blind, placebo-controlled, parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: Adult patients (>40 years old) 2 Possible or Probable Dementia associated with cerebrovascular disease as defined by NINDS-AIREN Criteria with dementia of greater than 3 months duration.

3. Radiological evidence of cerebrovascular disease. 4. Sex distribution: Both men and women. Women of child-bearing potential (<1 year post menopausal) must be willing to practice effective contraception and have a negative serum B-HCG at Screening. Pregnant and/or lactating females are excluded.

5. Race and Health: Any generally healthy, ambulatory or ambulatory aided (i.e., walker, cane or wheelchair) outpatient. Vision and hearing (glasses, contact lens, and hearing aid permissible), speech, motor function and comprehension must be sufficient for compliance with all testing procedures.

6. Patients with risk factors of hypertension and cardiac disease may be enrolled in the study, provided that hypertension is medication controlled (supine diastolic BP < 95 mm Hg) and cardiac disease (e.g. angina pectoris, congestive heart failure, right bundle branch block, or arrhythmias) is stable on appropriate medication for 3 months prior to Screening. Peripheral vascular disease must have been stable for 3 months prior to Screening. No elective surgical procedures should be planned during the course of the study (e.g., vascular bypass procedures or coronary artery bypass surgery).

7. Patients with risk factors of diabetes mellitus may be enrolled in the study, provided that the patient's disease is stable and that there have been no recent (within 3 months) admissions for diabetic ketoacidosis, hyperosmolar coma, or hypoglycemia. Patients with non-insulin-dependent diabetes may enroll in the study if controlled on diet or oral medications. All diabetic patients must have a HbA1c concentration of <=10% and a plasma glucose concentration of <= 250 mg/dL.

8. Patients with risk factors of stroke may be enrolled in the study, provided that the disease process has been stable or controlled on medication for greater than 3 months prior to Screening. Patients receiving anticoagulation with warfarin are eligible for inclusion in the study if the International Normalized Ratio (INR) for prothrombin time is within the therapeutic range for prophylaxis (1.4-3.0) and the dose of warfarin is stable.

-- Patients with prosthetic heart valves, who require full anticoagulation, should have a stable (>= 3 months) INR in the range of 2.5-3.5.

9. Patients who have taken a previously approved cholinesterase inhibitor (e.g., Aricept., Exelon., Reminyl., Cognex.) or memantine (Ebixa, Akinatol) are allowed provided that the medication was discontinued at least six (6) weeks prior to Screening.

10. Patients with thyroid disease may be included in the study, provided they are euthyroid on treatment.

11. Patient and study partner are willing to participate and have provided written Informed Consent prior to being exposed to any study-related procedures.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 974 (Actual)
Dates: Start 2003-03; Primary Completion 2005-08 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety: physical examinations, ECG and clinical laboratory tests. Efficacy: Vascular-Alzheimer's Disease Assessment Scale-Cognitive subscale (V-ADAS-cog) and the Clinician's Interview-Based Impression of Change-Plus Version (CIBIC-Plus). | Parameters will be measured prior to, during and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Posner, Study Director — Eisai Inc.
Locations (5):
- United States (5):
  - Central Arkansas Research (CARE), Hot Springs, Arkansas
  - Comprehensive Neuroscience, St. Petersburg, Florida
  - St. Francis Medical Center, Peoria, Illinois
  - Neurological Associate of Albany PC, Albany, New York
  - University of Texas Mental Sciences Institute, Houston, Texas